CLINICAL TRIAL: NCT04066244
Title: An Open-label, Adaptive Design Study in Patients With Amyotrophic Lateral Sclerosis (ALS) to Characterize Safety, Tolerability and Brain Microglia Response, as Measured by TSPO Binding, Following Multiple Doses of BLZ945 Using Positron Emission Tomography (PET) With the Radioligand [11C]-PBR28
Brief Title: Study of Safety and Proof of the Mechanism of BLZ945 in ALS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated after assessment of potential benefit-risk from available data
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBLZ945C12201; 2019-000826-22 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: PET; ALS; Microglia; CSF
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — 4-(2-(2-hydroxycyclohexylamino)benzothiazol-6-yloxy)pyridine-2-carboxylic acid methylamide

STUDY DESIGN:
Intervention Model Description: This study is an exploratory, adaptive, open-label study of single or multiple cycles of BLZ945 in participants with ALS. Cohorts 1-4 are not randomized, while Cohort 5 is randomized in open label two treatment arms. Cohorts 1-4 have single group design and Cohort 5 has parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Other): BLZ945 300mg
  Interventions: Drug: BLZ945
- Cohort 2 (Other): BLZ945 600mg
  Interventions: Drug: BLZ945
- Cohort 3 (Other): BLZ945 1200mg
  Interventions: Drug: BLZ945
- Cohort 4 (Other): BLZ945 800mg
  Interventions: Drug: BLZ945
- Cohort 5 Arm #1 (Other): BLZ945 800mg (4 days treatment + 10 days off)
  Interventions: Drug: BLZ945
- Cohort 5 Arm #2 (Other): BLZ945 800mg (once weekly)
  Interventions: Drug: BLZ945

INTERVENTIONS:
Drug: BLZ945 — Investigational drug capsules taken orally or via enteral infusion

SUMMARY:
It was an open label study to evaluate safety, tolerability and brain microglia response in participants with Amyotrophic Lateral Sclerosis (ALS) following multiple doses of BLZ945.

DETAILED DESCRIPTION:
The purpose of the study was to identify a dose (or doses) of BLZ945, that measurably decrease(s) 18 KDa Translocator Protein (TSPO) binding in the brain of participants with ALS. The study also aimed to evaluate the safety and tolerability of BLZ945 in participants with ALS at different doses and dosing regimens, and safety related effects on extracellular matrix (ECM) accumulation.

This was an exploratory, adaptive , open label study of approximately 16 participants in cohorts of 4 participants per cohort at increasing doses of BLZ945 with the last dose determined after the completion of cohorts 1 to 3.

Each cohort received treatment for 4 days and continued with a 32 day follow up period with an end of study visit at day 36.

After completion of the 4 initial cohorts a fifth cohort was initiated with two parallel arms receiving BLZ945 for up to 12 weeks at two different treatment regimens, either once weekly or 4 days of treatment followed by 10 days off drug.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate well with the investigator, to understand and comply with the study visits and procedures of the study
* Written informed consent must be obtained before any assessment is performed.
* Male and female participants who are 18 years old or older at screening, and who are diagnosed with familial or sporadic ALS according to the World Federation of Neurology Revised El Escorial criteria of either bulbar or limb onset.
* Disease duration from symptoms onset no longer than 48 months at the screening visit.
* Females of childbearing potential must have a negative pregnancy test at screening and/or baseline.
* Treatment with approved ALS therapies is allowed, but participants need to be on a stable dose and regimen for at least 30 days prior to baseline.
* Having completed the Core Treatment Period to be able to continue in the Extended Treatment Period.

Exclusion Criteria:

* A history of clinically significant ECG abnormalities
* Active medical or neurologic diseases other than ALS, that in the opinion of the investigator would limit their participation in the current study.
* Use of other investigational drugs within 5 half-lives of screening, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes.
* Presence of human immunodeficiency virus (HIV) infection based on screening lab results.
* Evidence of active or latent tuberculosis as assessed by Quantiferon testing at the screening visit.
* Positive serology for hepatitis B surface antigen, or hepatitis C antibodies confirmed by an appropriate licensed test at screening.
* Signs or symptoms, in the judgement of the investigator, of a clinically significant systemic viral, bacterial or fungal infection within 30 days prior to the screening visit.
* Cardiac disorders, such as recent cardiac history (within 6 months of screening) of acute coronary syndrome, acute heart failure, or significant ventricular arrhythmia at the screening visit or participants with a history of severe pulmonary hypertension. Participants with cardiac failure class 3 or 4 of the NYHA classification, or history of reduced LVEF or individuals with implanted cardiac pacemaker, or defibrillator.
* Significant hematological laboratory abnormalities.
* Clinical evidence of liver disease or liver injury or any of the following hepatic conditions at the screening visit:
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 14 days after last dose of BLZ945.
* Pregnant or nursing female participants
* Sexually active males unless they use a condom during intercourse while taking the drug during treatment, for 14 days after stopping BLZ945 and should not father a child in this period.
* History or presence of impaired renal function at the screening visit.
* Active suicidal ideation.
* History of drug abuse or harmful alcohol use within the 12 months prior to dosing within the judgement of the investigator, or evidence of such abuse as indicated by the laboratory assays conducted during screening.
* Active GI conditions such as Barrett's esophagus, achalasia, esophageal varices and active or history of esophageal cancer, pre-existing pancreatic disease at screening visit.
* History of active vasculitis or history of autoimmune disease autoimmune disease associated with vasculitis (eg., RA, SLE, Sjögrens disease, scleroderma).
* History or active cardiac valve disorder, congenital valve disease, or other clinical condition that might affect cardiac valve function
* Use of systemic anticoagulation that cannot be temporarily paused before study procedures
* Abnormal values on CT scan or echocardiography, signs of vasculitis, or evidence of a significant medical condition meeting treatment discontinuation criteria will be exclusionary for continuation in the extended treatment period.
* Participants who are planning to initiate treatment with an additional approved ALS therapy in the next 24 weeks are not allowed to continue in the extended treatment period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
- Novartis Investigative Site, Turku, Finland
- Novartis Investigative Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2560

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a screening and baseline period of up to 42 days for part 1 (Cohorts1-4) and of 6 weeks for part 2 (Cohort 5)
Groups:
- BLZ945 300mg - Cohort 1 (Part 1): BLZ945 300mg
- BLZ945 600mg - Cohort 2 (Part 1): BLZ945 600mg
- BLZ945 800mg - Cohort 4 (Part 1): BLZ945 800mg
- BLZ945 1200mg - Cohort 3 (Part 1): BLZ945 1200mg
- BLZ945 800mg - Cohort 5 Arm #1 (Part 2): BLZ945 800mg (4 days on/10 days off)
- BLZ945 800mg - Cohort 5 Arm #2 (Part 2): BLZ945 800mg (once weekly)
Period: Part 1 (Cohort 1-4)
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Started | 4 | 4 | 4 | 4 | 0 | 0
Completed | 4 | 4 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Cohort 5)
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Started | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 6 | 28
Age, Continuous [Median (Full Range); unit: years] | 50.5 [46 to 58] | 59.5 [33 to 76] | 65.5 [56 to 68] | 64 [62 to 68] | 55.5 [52 to 74] | 62.5 [32 to 67] | 60.5 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 1 | 2 | 10
  Male | 2 | 2 | 3 | 2 | 5 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 4 | 4 | 6 | 6 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1-4 : Change From Baseline in Volume of Distribution (Vt) in Different Brain Regions for [11C]-PBR28 PET Scan
Description: [11C]-PBR28 is a positron emission tomography (PET) radiotracer for the 18 kDa translocator protein (TSPO) that is used to image neuroinflammation in vivo. [11C]PBR28 imaging was used to measure microglial volume at baseline and after BLZ945 treatment in ALS participants.
  Relative % change from baseline in volume of distribution (Vt) of [11C]-PBR28 in different brain regions after BLZ945 treatment
Time Frame: Baseline, day 5
Population: PD analysis set, all participants in cohorts 1-4 with available PD data and no protocol deviations with relevant impact on PD data and with a valid assessment of the outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1)
Number analyzed (Participants) | 3 | 3 | 4 | 2
Percent change from baseline
  Precentral gyrus - day 5 | 0.67 (33.825) | -20.33 (16.458) | 9.90 (31.570) | -9.63 (1.516)
  Basal Ganglia - day 5 | -3.70 (22.729) | -15.18 (16.343) | 13.27 (35.504) | -10.73 (5.872)
  Brain Stem - day 5 | -7.10 (20.890) | -10.00 (13.464) | 50.56 (100.838) | -16.69 (61.674)
  Cerebellar White Matter - day 5 | -4.41 (20.678) | -14.11 (11.904) | 27.65 (60.112) | -16.87 (4.874)
  Cerebellum - day 5 | -3.53 (20.459) | -10.06 (8.365) | 17.52 (44.628) | -11.78 (3.854)
  Frontal Lobe - day 5 | 1.33 (30.101) | -18.67 (15.881) | 9.10 (29.745) | -9.70 (0.224)
  Occipital Lobe - day 5 | -3.01 (23.217) | -11.50 (10.457) | 14.18 (36.595) | -5.87 (0.292)
  Thalamus - day 5 | -8.00 (22.581) | -14.85 (13.466) | 13.89 (42.938) | -14.14 (3.521)
  Whole Brain - day 5 | -0.95 (26.606) | -15.59 (14.716) | 12.22 (34.922) | -7.72 (0.326)

2. Primary Outcome: Cohort 5 (PET Sub-study): Change From Baseline in Volume of Distribution (Vt) in Different Brain Regions for [11C]-PBR28 PET Scan
Description: as for outcome 1
Time Frame: Baseline, day 84
Population: PD analysis set, all participants in cohort 5 with available PD data and no protocol deviations with relevant impact on PD data and with a valid assessment of the outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 1 | 0
Percent change from baseline
  Precentral gyrus - day 84 | -21.95 |
  Basal Ganglia - day 84 | -17.80 |
  Brain Stem - day 84 | -26.10 |
  Cerebellar White Matter - day 84 | -22.40 |
  Cerebellum - day 84 | -19.40 |
  Frontal Lobe - day 84 | -21.53 |
  Occipital Lobe - day 84 | -17.76 |
  Thalamus - day 84 | -29.39 |
  Whole Brain - day 84 | -20.51 |

3. Primary Outcome: Cohort 5: Change From Baseline in Esophageal Wall Thickness
Description: Mean change from baseline in esophageal wall thickness measured in mm
Time Frame: Baseline, Day 84
Population: Full analysis set, participants in cohort 5 that received any study drug with a valid assessment for the outcome measure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 4 | 2
mm
  Wall thickness average: number analyzed (Participants) | 2 | 2
  Wall thickness average | 0.258 (0.7990) | 0.758 (2.1708)
  Lower third Wall Thickness: number analyzed (Participants) | 2 | 2
  Lower third Wall Thickness | 0.040 (0.9475) | -1.400 (2.9981)
  Middle third Wall Thickness: number analyzed (Participants) | 2 | 2
  Middle third Wall Thickness | 0.235 (0.0212) | 2.795 (2.6234)
  Upper third Wall Thickness: number analyzed (Participants) | 2 | 2
  Upper third Wall Thickness | 0.500 (1.4284) | 0.880 (0.8910)

4. Primary Outcome: Cohort 5: Cardiac Valve Thickness at Day 84 Compared to Baseline
Description: Cardiac valve thickness on a three point ordinal scale. Categorized by imaging vendor into three semiquantitative (normal, mild-moderate and severe) categories
Time Frame: Baseline, Day 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 6 | 6
Participants
  Aortic valve thickness - Baseline: Normal | 6 | 6
  Aortic valve thickness - Baseline: Mild- Moderate | 0 | 0
  Aortic valve thickness - Day 84: number analyzed (Participants) | 2 | 2
  Aortic valve thickness - Day 84: Normal | 2 | 2
  Aortic valve thickness - Day 84: Mild- Moderate | 0 | 0
  Mitral valve thickness - Baseline: Normal | 6 | 5
  Mitral valve thickness - Baseline: Mild- Moderate | 0 | 1
  Mitral valve thickness - Day 84: number analyzed (Participants) | 2 | 2
  Mitral valve thickness - Day 84: Normal | 2 | 2
  Mitral valve thickness - Day 84: Mild- Moderate | 0 | 0
  Pulmonary valve thickness - Baseline: Normal | 6 | 6
  Pulmonary valve thickness - Baseline: Mild- Moderate | 0 | 0
  Pulmonary valve thickness - Day 84: number analyzed (Participants) | 2 | 2
  Pulmonary valve thickness - Day 84: Normal | 2 | 2
  Pulmonary valve thickness - Day 84: Mild- Moderate | 0 | 0
  Tricuspid valve thickness - Baseline: Normal | 6 | 6
  Tricuspid valve thickness - Baseline: Mild- Moderate | 0 | 0
  Tricuspid valve thickness - Day 84: number analyzed (Participants) | 2 | 2
  Tricuspid valve thickness - Day 84: Normal | 2 | 2
  Tricuspid valve thickness - Day 84: Mild- Moderate | 0 | 0

5. Primary Outcome: Cohort 5: Cardiac Valve Stenosis at Day 84 Compared to Baseline
Description: Cardiac valve stenosis on a four point ordinal scale. Categorized by imaging vendor into four semiquantitative (normal, mild, moderate and severe) categories
Time Frame: Baseline, Day 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 6 | 6
Participants
  Aortic valve - Baseline: Normal | 6 | 6
  Aortic valve - Baseline: Mild | 0 | 0
  Aortic valve - Day 84: number analyzed (Participants) | 2 | 2
  Aortic valve - Day 84: Normal | 2 | 2
  Aortic valve - Day 84: Mild | 0 | 0
  Mitral valve - Baseline: Normal | 6 | 6
  Mitral valve - Baseline: Mild | 0 | 0
  Mitral valve - Day 84: number analyzed (Participants) | 2 | 2
  Mitral valve - Day 84: Normal | 2 | 2
  Mitral valve - Day 84: Mild | 0 | 0
  Pulmonary valve - Baseline: Normal | 6 | 6
  Pulmonary valve - Baseline: Mild | 0 | 0
  Pulmonary valve thickness - Day 84: number analyzed (Participants) | 2 | 2
  Pulmonary valve thickness - Day 84: Normal | 2 | 2
  Pulmonary valve thickness - Day 84: Mild | 0 | 0
  Tricuspid valve - Baseline: Normal | 6 | 6
  Tricuspid valve - Baseline: Mild | 0 | 0
  Tricuspid valve - Day 84: number analyzed (Participants) | 2 | 2
  Tricuspid valve - Day 84: Normal | 2 | 2
  Tricuspid valve - Day 84: Mild | 0 | 0

6. Primary Outcome: Cohort 5: Cardiac Valve Regurgitation Severity at Day 84 Compared to Baseline
Description: Cardiac valve regurgitation severity on a four point ordinal scale. Categorized by imaging vendor into four semiquantitative (normal, mild, moderate and severe) categories
Time Frame: Baseline, Day 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 6 | 6
Participants
  Aortic valve - Baseline: Normal | 5 | 6
  Aortic valve - Baseline: Mild | 1 | 0
  Aortic valve - Day 84: number analyzed (Participants) | 2 | 2
  Aortic valve - Day 84: Normal | 2 | 2
  Aortic valve - Day 84: Mild | 0 | 0
  Mitral valve - Baseline: Normal | 3 | 3
  Mitral valve - Baseline: Mild | 3 | 3
  Mitral valve - Day 84: number analyzed (Participants) | 2 | 2
  Mitral valve - Day 84: Normal | 0 | 1
  Mitral valve - Day 84: Mild | 2 | 1
  Pulmonary valve - Baseline: Normal | 3 | 4
  Pulmonary valve - Baseline: Mild | 3 | 2
  Pulmonary valve - Day 84: number analyzed (Participants) | 2 | 2
  Pulmonary valve - Day 84: Normal | 2 | 1
  Pulmonary valve - Day 84: Mild | 0 | 01
  Tricuspid valve - Baseline: Normal | 3 | 2
  Tricuspid valve - Baseline: Mild | 3 | 4
  Tricuspid valve - Day 84: number analyzed (Participants) | 2 | 2
  Tricuspid valve - Day 84: Normal | 1 | 1
  Tricuspid valve - Day 84: Mild | 1 | 1

7. Primary Outcome: Cohort 5: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Mean change from baseline in Left Ventricular Ejection Fraction.
  LVEF is defined as the percentage of blood volume ejected from the left ventricle during systole (contraction phase) relative to the total volume of blood present in the ventricle at the end of diastole (relaxation phase).
Time Frame: Baseline, day 84
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 2 | 2
Percentage of LVEF | 1.533 (2.9713) | 5.021 (2.0796)

8. Primary Outcome: Cohort 5: Adverse Events Related to Extracellular Matrix (ECM) Accumulation
Description: Number of patients with adverse events related to ECM accumulation
Time Frame: Up to Day 84
Population: Full analysis set, participants in cohort 5 that received any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 6 | 6
Participants | 2 | 2

9. Secondary Outcome: Cohorts 1-5: Plasma Pharmacokinetics (PK) of BLZ945 - Cmax
Description: Measured by Cmax - The maximum plasma concentration of BLZ945
Time Frame: Cohort 1-4: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours after BLZ945 dosing on Day 1 and Day 4. Cohort 5: pre-dose, 1, 2 and 4 hours after BLZ945 dosing on Day 1 (Arm#2 only) and Day 4 (Arm#1 only)
Population: Participants in the PK analysis set with an available value for the outcome measure at the corresponding timepoint.
  The PK analysis set included all participants with at least one available valid PK concentration measurement, who received any study drug, and had no protocol deviations that impacted on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL of BLZ945
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 6
ng/mL of BLZ945
  Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3 | 0 | 6
  Day 1 | 6850 (780) | 16000 (2510) | 21100 (5630) | 25900 (2630) |  | 19900 (5990)
  Day 4: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 0
  Day 4 | 12100 (2300) | 25900 (3440) | 30700 (7800) | 37600 (4270) | 22400 (3120) |

10. Secondary Outcome: Cohorts 1-5: Plasma Pharmacokinetics (PK) of BLZ945 - Tmax
Description: Measured by Tmax - Time to Reach the Maximum Concentration After Drug Administration of BLZ945.
  Actual recorded sampling times were taken into consideration for the calculation of PK parameters.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 6
hours
  Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3 | 0 | 6
  Day 1 | 1.02 [1.00 to 1.07] | 2.01 [1.00 to 2.08] | 2.01 [1.00 to 7.00] | 1.00 [1.00 to 1.00] |  | 2.00 [1.00 to 4.17]
  Day 4: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 0
  Day 4 | 1.01 [0.500 to 1.03] | 1.50 [1.00 to 4.00] | 3.00 [1.00 to 6.08] | 2.02 [1.00 to 4.00] | 1.49 [0.817 to 2.00] |

11. Secondary Outcome: Cohorts 1-5: Plasma Pharmacokinetics (PK) of BLZ945 - AUC
Description: Measured by AUC - Area under the curve of BLZ945
  AUC0-24h is the AUC calculated from time zero to 24 hours after dosing (end of a dosing interval).
  AUClast is the AUC from time zero to the last measurable concentration sampling time.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour * ng/mL
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 6
hour * ng/mL
  AUC 0-24h - Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3 | 0 | 0
  AUC 0-24h - Day 1 | 93000 (2510) | 204000 (28000) | 278000 (49600) | 391000 (10600) |  |
  AUC 0-24h - Day 4: number analyzed (Participants) | 4 | 4 | 4 | 3 | 0 | 0
  AUC 0-24h - Day 4 | 175000 (14100) | 401000 (88700) | 535000 (157000) | 680000 (48300) |  |
  AUClast - Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3 | 0 | 6
  AUClast - Day 1 | 92600 (2750) | 203000 (26800) | 277000 (99500) | 34100 (91100) |  | 56900 (21400)
  AUClast - Day 4: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 0
  AUClast - Day 4 | 170000 (20300) | 399000 (87800) | 533000 (158000) | 671000 (43400) | 73400 (7710) |

12. Secondary Outcome: Cohorts 1-4: Plasma Pharmacokinetics (PK) of BLZ945 - T1/2
Description: Measured by T1/2 - The elimination half-life of BLZ945
Time Frame: Cohort 1-4: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours after BLZ945 dosing on Day 1 and Day 4.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1)
Number analyzed (Participants) | 4 | 4 | 4 | 3
Hours
  Day 1 | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75.
  Day 4 | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75. | NA (NA) — Not estimable because the R-squared of the terminal elimination phase was less than 0.75.

13. Secondary Outcome: Cohorts 1-4: Renal Clearance (CLR) of BLZ945
Description: Urine renal clearance (CLR) of BLZ945
Time Frame: pre-dose, 0-4, 4-8, 8-12 and 12-24 hours after BLZ945 dosing on Day 1 and Day 4
Population: PK analysis set, participants with at least one available valid PK concentration measurement , who received any study drug, and had no protocol deviations that impact on PK data
Measure: Mean (Standard Deviation); unit: liter/hour (L/hr)
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1)
Number analyzed (Participants) | 4 | 4 | 4 | 3
liter/hour (L/hr)
  Day 1: number analyzed (Participants) | 4 | 4 | 3 | 3
  Day 1 | 0.00597 (0.00184) | 0.00844 (0.00675) | 0.00466 (0.00312) | 0.0213 (0.0258)
  Day 4: number analyzed (Participants) | 4 | 3 | 4 | 2
  Day 4 | 0.00667 (0.00127) | 0.00410 (0.00205) | 0.00362 (0.00262) | 0.00550 (0.00129)

14. Secondary Outcome: Cohorts 1-5: Number of Patients With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence and severity of AEs and SAEs by treatment group.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5. For CTCAE, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE
Time Frame: From first dose of study treatment up to 32 days after last dose (Day 36) for Cohorts 1-4 and up to 4 weeks after last dose (Day 330) for Cohort 5. *Maximum duration of exposure in Cohort 5 was 302 days. 302 + 28 days of FU=330 days
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BLZ945 300mg - Cohort 1 (Part 1) | BLZ945 600mg - Cohort 2 (Part 1) | BLZ945 1200mg - Cohort 3 (Part 1) | BLZ945 800mg - Cohort 4 (Part 1) | BLZ945 800mg - Cohort 5 Arm #1 (Part 2) | BLZ945 800mg - Cohort 5 Arm #2 (Part 2)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 6
Participants
  Total AEs | 2 | 2 | 4 | 4 | 6 | 6
  AE of grade 1 | 2 | 2 | 4 | 4 | 5 | 6
  AE of grade 2 | 2 | 1 | 2 | 3 | 5 | 5
  AE of grade 3 | 0 | 0 | 0 | 2 | 1 | 5
  AE of grade 4 | 0 | 0 | 0 | 0 | 0 | 1
  AE of grade 5 | 0 | 0 | 0 | 0 | 0 | 2
  Study drug-related AEs | 2 | 2 | 2 | 3 | 5 | 5
  Serious AEs | 0 | 0 | 0 | 1 | 0 | 4
  AEs leading to discontinuation of study treatment | 0 | 0 | 0 | 0 | 0 | 4
  Study-drug related AEs leading to discontinuation of study treatment | 0 | 0 | 0 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 32 days after last dose (Day 36) for Cohorts 1-4 and up to 4 weeks after last dose (Day 330) for Cohort 5. *Maximum duration of exposure in Cohort 5 was 302 days. 302 + 28 days of FU=330 days
Groups:
- BLZ945 300mg: BLZ945 300mg
- BLZ945 600mg: BLZ945 600mg
- BLZ945 800mg: BLZ945 800mg
- BLZ945 1200mg: BLZ945 1200mg
- Arm 1 (4/10): Arm 1 (4/10)
- Arm 2 (4/10) QW: Arm 2 (4/10) QW
- Total: Total
Arm/Group | BLZ945 300mg | BLZ945 600mg | BLZ945 800mg | BLZ945 1200mg | Arm 1 (4/10) | Arm 2 (4/10) QW | Total
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 2/6 | 2/28
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 1/4 | 0/6 | 4/6 | 5/28
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 4/4 | 4/4 | 6/6 | 6/6 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BLZ945 300mg (N=4) | BLZ945 600mg (N=4) | BLZ945 800mg (N=4) | BLZ945 1200mg (N=4) | Arm 1 (4/10) (N=6) | Arm 2 (4/10) QW (N=6) | Total (N=28)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BLZ945 300mg (N=4) | BLZ945 600mg (N=4) | BLZ945 800mg (N=4) | BLZ945 1200mg (N=4) | Arm 1 (4/10) (N=6) | Arm 2 (4/10) QW (N=6) | Total (N=28)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 3 | 1 | 9
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 2 | 3 | 2 | 8
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 2 | 5
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Faecal volume decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 1 | 1 | 7
Headache (Nervous system disorders) | 2 | 0 | 0 | 3 | 3 | 2 | 10
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT04066244/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT04066244/SAP_001.pdf